CLINICAL TRIAL: NCT05198271
Title: Effect of Controlling Environmental Risk Factors in Established RA
Acronym: DISRUPT-estRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL21_0533
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: prevention; smoking; diet; periodontitis; physical activity; stress
MeSH Terms: conditions — Arthritis, Rheumatoid; Smoking; Periodontitis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Management of risk factors (Experimental): -6 month program for reduction /correction of risk factors in patient with active RA :
  1. Smoking cessation
  2. weightloss
  3. Increased physical activity
  4. Periodontal treatment
  5. Decreased anxiety
  Interventions: Other: Management of risk factors; Behavioral: Smoking cessation; Behavioral: weightloss; Other: periodontal disease treatment; Behavioral: increased physical activity; Behavioral: Decreased anxiety

INTERVENTIONS:
Other: Management of risk factors — * For all patients:
    * Online dietician consultation (45 min 1st consultation with set objectives then 15-20 min for the following ones) then proposal of varied weekly menus, adapted to different cultural and social contexts by email and reassessment at M3 and M6
    * Clinical and radiographic periodontological evaluation at M0 and M6 by a specialist with dental hygiene advice with delivery of equipment and scaling
    * Initial teleconsultation with motivational interview by sports doctor / APA (30 min) with evaluation of initial physical activity, search for contraindications and development of a personalized program with aerobic and resistance training. Provision of filmed sessions and digital exercise materials for regular practice at home and self-assessment using data from the accelerometer with automatic online report.
  * Motivational supports on the MyGoodLife / MyGoodCare platform (weight, food questionnaire, pedometer, tobacco consumption)
Behavioral: Smoking cessation — - For active smoking patients:
  * Tobacco consultations: S0, S4 and S8 then according to the opinion of the tobacco specialist
  * Nicotine substitutes +/- varenicline according to tobacco consumption
  * Online notebook to record tobacco consumption and "triggers"
Behavioral: weightloss — -For overweight or obese patients: Online dietician consultation every 15 days for 3 months, the consultation based on the online filling of food questionnaires and the weight curve
Other: periodontal disease treatment — - For patients with periodontal disease: treatment of periodontal disease (planing, cast splint, tooth avulsion, etc.) between M0 and M3, dental panoramic M0 at inclusion and M6
Behavioral: increased physical activity — - For patients with low physical activity: Follow-up by level gp session: 45 '/ week for 3 months
Behavioral: Decreased anxiety — - For anxious patients:
  * Teleconsultation with a psychiatrist specializing in stress management, global assessment, identification of the factors involved and training in the use of cardiac coherence
  * Delivery of connected equipment for the practice of cardiac coherence

SUMMARY:
* The factors contributing to the development of rheumatoid arthritis are multiple, with a role of the environment and a predisposing genetic background.
* Among the modifiable environmental factors :unbalanced diet, overweight, low physical activity, smoking, periodontal disease, stress have been identified as risk factors for developing RA.
* By causing low-grade inflammation and stimulation of the immune system (particularly through adipokines, citrullination phenomena and changes in the microbiota), these factors promote the onset of the disease and could also participate in the maintenance of inflammatory processes.
* Thus, obese subjects have more active RA, a lower therapeutic response, and weight loss is associated with lower disease activity ; sedentary lifestyle is associated with more active RA and increased physical activity has beneficial effects on RA; people who smoke respond less well to treatment; periodontal disease is associated with more active RA and their treatment is associated with a decrease in this activity.
* Finally, different methods having a beneficial impact on stress (mindfulness meditation, yoga, relaxation, etc.) have shown interesting results in patients with RA.
* It is important to note that all of these factors are also associated with an increased cardiovascular risk, the leading cause of death in RA.
* The combination of these factors probably has synergistic effects and it is therefore relevant to propose a correction of all these factors in the same program.
* We have developed a management program for environmental risk factors for RA based with experts including rheumatologists, nutritionists, smoking cessation specialists, periodontal disease specialists and stress specialists.

DETAILED DESCRIPTION:
Methodology:

* We will conduct a Phase 2 to one phase trial with A'Hern design.
* The patients included will have RA (ACR / EULAR 2010 criteria), with an active disease (2.6 <DAS 28 <5.1), and at least 3 risk factors among: BMI ≥25 kg / m², low physical activity , active smoking, periodontitis and anxiety.

  1. The primary endpoint will be the number of patients for whom at least 2 or 3 risk factors (depending on whether 3 present or 4-5 present at baseline) are corrected / in the process of being corrected at 6 months.
  2. The secondary endpoints will be:

A) Acceptability: number of patients agreeing to participate in the protocol / total number of screened patients fulfilling the inclusion criteria; questionnaires with EVA carried out at the end of the program; Membership of the program: online completion of questionnaires, use of the accelerometer, participation in teleconsultations and organized group sessions.

B) For each risk factors: number of patients who corrected it at 3 and 6 months.

C) RA activity measured by DAS28-CRP + RAID questionnaire, biological markers

D) Distribution of the different germs of the oral and faecal micobiota and diversity.

* As risks factor are established chronically, we hypothesize that only 10% of patients would correct at least 2 or 3 risk factors over 6 months in the absence of intervention. The expected efficiency is 40%.
* By recruiting 25 patients, we will have a power of 90% to demonstrate that the one-sided 95% confidence interval of the effectiveness of the intervention is greater than 10% (p (0) if the true value of effectiveness is 35% (p (1)). This demonstration will be made if 6 patients out of 25 are successful.

Procedure:

* 3 visits will be necessary for rheumatological and biological evaluations (inclusion +/- M0, M3 and M6).
* All patients will have 2 periodontal visits (M0 and M6 for evaluation and scaling). Those with periodontitis will have other visits depending on the care to be performed.
* The smoking patients will have teleconsultations (TC) with a tobacco specialist (S0, S4 and S8 then according to tobacco specialist).
* All patients will have a TC with a dietitian (45 min 1st consultation with set goals) and those overweight will then have a TC every 15 days for 3 months.
* All patients will have a TC with a sports doctor (assessment of physical activity and development of a personalized program, explanation of the pedometer provided). For those with low physical activity, a virtual group session of 45 min / week will be organized.
* Patients with anxiety will have TC with a psychiatrist specializing in stress management, with training in the use of cardiac coherence from connected equipment given to the patient.
* All the interventions will be coordinated on an existing platform (MyGoodLife) which allows the dietary assessment, the automatic report of connected objects (pedometer) and the organization of group sessions.

ELIGIBILITY:
Inclusion Criteria:

* RA (ACR / EULAR 2010 criteria), with an active disease (2.6 <DAS 28 <5.1)
* Basis treatment for at least 3 months and corticoids <= 10mg / day

And at least 3 risk factors among:

* BMI ≥25 kg / m²
* Low physical activity (IPAQ short version)
* Active smoking
* Periodontitis ( bone loss on dental panoramic)
* Anxiety ( Beck anxiety Index > 16)

Exclusion Criteria:

* Patient under protective measure or unable to consent
* Patient for whom a change in basic treatment for RA is planned within 6 months
* Active cancer
* Active infection
* Antibiotic therapy in the previous 3 months
* No health cover
* Diabetes
* Unbalanced psychiatric pathologies
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the effectiveness at 6 months of this program on the overall reduction / correction of risk factors. | 6 MONTHS
  Number of patients for whom at least 2 or 3 risk factors (depending on whether 3 present or 4-5 present at baseline) are corrected / in the process of correction.
  Risk factors will be considered corrected / in the process of being corrected if:
  * Weight loss ≥5% of initial weight at 6 months (objective measurement of weight) and / or BMI at 6 months < 25kg/m²
  * Complete smoking cessation (declarative assessment)
  * Correction of sedentary lifestyle with moderate to strong IPAQ AND increase of ≥2,000 steps / day compared to the initial assessment (on average 5 days / 7) (questionnaire and quantified assessment obtained with the pedometer and automatically reported on the platform)
  * Improvement in periodontal disease scores ≥4 points on 6 teeth assessed according to Ramfjord's recommendation (plaque index (Sillness and Loe index), gingival (Lobene index) and papillary bleeding index) (evaluation by the periodontologist)
  * Decrease in anxiety score from N class to N-1 class

SECONDARY OUTCOMES:
To assess the acceptability and adherence of RA patients to the intervention program. | 6 MONTHS
  * Acceptability:
    * number of patients agreeing to participate in the protocol / total number of screened patients fulfilling the inclusion criteria.
    * questionnaire with different visual analog scales carried out at the end of the program.
  * Adherence: assessed by completing online questionnaires / weight, using the accelerometer, participating in various teleconsultations and organized group sessions
At least two risk factors (if 3 present at base) or at least three (if 4 or 5 present at base) are corrected / in the process of correction. | 3 MONTHS
  same description as for the outcome 1
RA activity | 3 MONTHS, 6 MONTHS
  DAS 28-CRP, RAID, biological markers (FR, ACPA, CRP)
Distribution of the different germs of the oral and fecal micobiota and alpha and beta diversity | 3 MONTHS, 6 MONTHS
  targeted metagenomics 16s RNA
Personality traits assessed by the Minnesota Multiphasic Personality Inventory questionnaire (MMPI) | MONTH 0

CONTACTS AND LOCATIONS:
Overall Officials: Claire DAIEN, MD, Study Director — UH of Montpellier
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided